CLINICAL TRIAL: NCT00373217
Title: Evaluation of the Immunogenicity of Vaccination With Synthetic Peptides in Adjuvant in Patients With Advanced Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Brief Title: Vaccine Therapy, Paclitaxel, and Carboplatin in Treating Patients Who Are Undergoing Surgery for Stage III or Stage IV Ovarian Cancer, Primary Peritoneal Cancer, or Fallopian Tube Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment rate.
Sponsor: Craig L Slingluff, Jr (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Craig L Slingluff, Jr, Professor of Surgery, University of Virginia
Organization: University of Virginia (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10134; UVACC-OVA-2; UVACC-PRC-236-02
Record Dates: First submitted 2006-09-06; First posted 2006-09-07 (Estimated); Results first posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-08

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: fallopian tube cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — MAGEA1 protein, human; Receptor Protein-Tyrosine Kinases; Carboplatin; Paclitaxel

ARMS (2):
- Group 1 (Experimental): Patients in group one will receive a 3-hour infusion of paclitaxel and an infusion of carboplatin in week 1. Treatment may repeat every 3 weeks for up to four courses. They will then undergo surgery to remove as much of the tumor as possible. Within 2 weeks after surgery, patients will receive an injection of the vaccine once a week for 3 weeks. Treatment may repeat every 14 weeks for two courses. After finishing the first course of vaccine therapy, patients will receive a 3-hour infusion of paclitaxel and an infusion of carboplatin every 3 weeks for up to four courses.
  Interventions: Biological: MAGE-A1, Her-2/neu, FBP peptides ovarian cancer vaccine; Biological: tetanus toxoid helper peptide; Drug: carboplatin; Drug: paclitaxel; Procedure: conventional surgery
- Group 2 (Experimental): Patients in group two will undergo surgery to remove as much of the tumor as possible. Within 2 weeks after surgery, patients will receive an injection of the vaccine once a week for 3 weeks. Treatment may repeat every 14 weeks for two courses. After finishing the first course of vaccine therapy, patients will receive a 3-hour infusion of paclitaxel and an infusion of carboplatin every 3 weeks for up to eight courses. Some patients may undergo a second surgery within 6 weeks after completing the fourth course of chemotherapy and undergo tumor and/or lymph node tissue collection.
  Interventions: Biological: MAGE-A1, Her-2/neu, FBP peptides ovarian cancer vaccine; Biological: tetanus toxoid helper peptide; Drug: carboplatin; Drug: paclitaxel; Procedure: conventional surgery

INTERVENTIONS:
Biological: MAGE-A1, Her-2/neu, FBP peptides ovarian cancer vaccine — Given intradermally or subcutaneously
Biological: tetanus toxoid helper peptide — Given intradermally or subcutaneously
Drug: carboplatin — Given IV
Drug: paclitaxel — Given IV
Procedure: conventional surgery — Patients undergo primary optimal cytoreductive surgery

SUMMARY:
RATIONALE: Vaccines made from peptides may help the body build an effective immune response to kill tumor cells. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving vaccine therapy and chemotherapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well giving vaccine therapy together with paclitaxel and carboplatin works in treating patients who are undergoing surgery for stage III or stage IV ovarian cancer, primary peritoneal cancer, or fallopian tube cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the immunogenicity of vaccine therapy comprising synthetic ovarian cancer-associated peptides administered with a synthetic tetanus toxoid helper peptide emulsified in Montanide ISA-51 before or after paclitaxel and carboplatin in patients with stage III-IV ovarian epithelial, primary peritoneal cavity, or fallopian tube cancer undergoing optimal cytoreductive surgery.

OUTLINE: This is an open-label study. Patients are assigned to 1 of 2 treatment groups.

* Group 1:

  * Neoadjuvant chemotherapy:Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients then proceed to surgical debulking.
  * Surgical debulking: Patients undergo primary optimal cytoreductive surgery.
  * Vaccine therapy: Within 14 days after surgery, patients receive vaccine therapy comprising synthetic ovarian cancer-associated peptides, MAGE-A1:161-169, FBP:1901-199, Her-2/neu:369-377, MAGE-A1:96-104, and Her-2/neu:754-762, and tetanus toxoid helper peptide emulsified in Montanide ISA-51 intradermally and subcutaneously on days 1, 8, and 15. Treatment repeats every 14 weeks for 2 courses.
  * Adjuvant chemotherapy: Patients receive 4 courses of paclitaxel and carboplatin as in neoadjuvant chemotherapy after completion of course 1 of vaccine therapy.
* Group 2:

  * Surgical debulking: Patients undergo up-front optimal cytoreductive surgery. Patients with non-optimal primary debulking may undergo interval debulking surgery within 6 weeks after completing course 4 of adjuvant chemotherapy. If interval debulking surgery is performed, tumor and/or lymph node tissue is collected.
  * Vaccine therapy: Patients receive 2 courses of vaccine therapy as in group 1.
  * Adjuvant chemotherapy: Patients receive paclitaxel and carboplatin as in group 1, neoadjuvant chemotherapy. Treatment repeats every 21 days for up to 8 courses.

Patients undergo periodic blood and tumor tissue collection during study for correlative immunological analysis.

After completion of study treatment, patients with progressive disease are followed at 30 days and then every six months thereafter. All other patients are followed every 3 months for 36 months until disease progression or until another therapy is initiated, and then every six months thereafter.

PROJECTED ACCRUAL: A total of 28 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of ovarian epithelial, primary peritoneal cavity, or fallopian tube cancer

  * Stage III or IV disease
* HLA-A1, -A2, and/or -A3 positive
* Must have at least 1 undissected axillary or inguinal lymph node basin
* No recurrent disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Hemoglobin ≥ 8.0 g/dL
* WBC > 3,000/mm^3
* Absolute neutrophil count > 1,500/mm^3
* Hemoglobin A1c < 7%
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN
* HIV negative
* Hepatitis C negative
* No known or suspected allergies to any component of the study vaccine
* No other concurrent malignancy (except for nonmelanoma skin cancer) unless the patient was curatively treated and has been disease free for ≥ 5 years
* No active serious infection
* No autoimmune disorder with visceral involvement
* No prior or active autoimmune disorders requiring cytotoxic or immunosuppressive therapy

  * The following immunologic conditions are allowed:

    * Laboratory evidence of autoimmune disease (e.g., positive antinuclear antibody titer) without symptoms
    * Clinical evidence of vitiligo
    * Other forms of depigmenting illness
    * Mild arthritis requiring NSAIDs
* No New York Heart Association class III or IV heart disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No medical contraindication or potential problem that would preclude study compliance

PRIOR CONCURRENT THERAPY:

* At least 2 weeks since prior and no other concurrent chemotherapy, radiotherapy, or immunotherapy (e.g., interferons, tumor necrosis factor, interleukins, or monoclonal antibodies)
* More than 4 weeks since prior and no other concurrent investigational agents
* More than 4 weeks since prior and no concurrent allergy desensitization injections
* More than 4 weeks since prior and no concurrent oral or parenteral systemic corticosteroids
* No prior or concurrent inhaled corticosteroids (e.g., fluticasone and salmetrol, fluticasone, or triamcinolone acetonide)

  * Prior or concurrent topical corticosteroids allowed
* No prior vaccination with MAGE-A1:161-169, FBP:1901-199, Her-2/neu:369-377, MAGE-A1:96-104, or Her-2/neu:754-762
* More than 4 weeks since prior and no concurrent growth factors (e.g., epoetin alfa, darbepoetin alfa, or pegfilgrastim)
* No concurrent treatment for recurrent disease
* No concurrent nitrosoureas
* No concurrent illegal drug use
* Concurrent nonsteroidal anti-inflammatory drugs (NSAIDs), antihistamines, and chronic medications, unless excluded, are allowed
* Short-term therapy for acute conditions not specifically related to ovarian cancer is allowed

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-04-13 (Actual); Primary Completion 2008-02-07 (Actual); Study Completion 2008-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig L Slingluff, MD, Study Director — University of Virginia
Locations (1):
- University of Virginia Cancer Center, Charlottesville, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Adjuvant: Patients in group one will receive a 3-hour infusion of paclitaxel and an infusion of carboplatin in week 1. Treatment may repeat every 3 weeks for up to four courses. They will then undergo surgery to remove as much of the tumor as possible. Within 2 weeks after surgery, patients will receive an injection of the vaccine once a week for 3 weeks. Chemotherapy may repeat every 14 weeks for two courses. After finishing the first course of vaccine therapy, patients will receive a 3-hour infusion of paclitaxel and an infusion of carboplatin every 3 weeks for up to four courses.
  MAGE-A1, Her-2/neu, FBP peptides ovarian cancer vaccine: Given intradermally or subcutaneously
  tetanus toxoid helper peptide: Given intradermally or subcutaneously
  carboplatin: Given IV
  paclitaxel: Given IV
  conventional surgery: Patients undergo primary optimal cytoreductive surgery
  Vaccines are administered after chemotherapy and surgery, on weeks 0, 1, 2. Carboplatin and paclitaxel are administered weeks 3-24, then 3 more vaccines are administered week 23-25.
- Group 2: Neoadjuvant: Patients in group two will undergo surgery to remove as much of the tumor as possible. Within 2 weeks after surgery, patients will receive an injection of the vaccine once a week for 3 weeks. Treatment may repeat every 14 weeks for two courses. After finishing the first course of vaccine therapy, patients will receive a 3-hour infusion of paclitaxel and an infusion of carboplatin every 3 weeks for up to eight courses. Some patients may undergo a second surgery within 6 weeks after completing the fourth course of chemotherapy and undergo tumor and/or lymph node tissue collection.
  MAGE-A1, Her-2/neu, FBP peptides ovarian cancer vaccine: Given intradermally or subcutaneously
  tetanus toxoid helper peptide: Given intradermally or subcutaneously
  carboplatin: Given IV
  paclitaxel: Given IV
  conventional surgery: Patients undergo primary optimal cytoreductive surgery
  Vaccines are administered after surgery, on weeks 0, 1, 2. Carboplatin and paclitaxel are administered weeks 3-12, then 3 more vaccines are administered week 14-16.
Period: Overall Study
Arm/Group | Group 1: Adjuvant | Group 2: Neoadjuvant
Started | 3 | 3
Completed | 2 | 3
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 56.4 [49.4 to 68.9] | 53.9 [49.9 to 56.2] | 55.2 [49.4 to 68.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cytotoxic T-cell Response to Vaccine Therapy Comprising 5 Synthetic Ovarian Cancer-associated Peptides, as Assessed Using Peripheral Blood During Course 1
Description: T cell response by interferon-gamma ELIspot assay, after 1 in vitro stimulation
Time Frame: through week 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Adjuvant | Group 2: Neoadjuvant
Number analyzed (Participants) | 3 | 3
Participants | 1 | 1

2. Secondary Outcome: Cytotoxic T-cell Response to Vaccine Therapy Comprising Synthetic Ovarian Cancer-associated Peptides, as Assessed Using Peripheral Blood During Chemotherapy and During Course 2
Description: T cell response to one or more peptides in peripheral blood by IFN-gamma ELIspot assay during chemotherapy and/or during 2nd course of vaccines.
Time Frame: weeks 4-28 for group 1, week 4-16 for group 2
Population: Participants evaluated for immune response during chemotherapy and/or during vaccine course 2. One participant in adjuvant arm (1) came off study after week 3 and was not evaluable for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Adjuvant | Group 2: Neoadjuvant
Number analyzed (Participants) | 2 | 3
Participants | 2 | 1

3. Secondary Outcome: Cytotoxic T-cell Response Against Autologous and/or Major Histocompatibility Complex-matched Allogeneic Tumor Cells Pre- and Post-treatment
Description: T cell responses to tumor cells in vitro. Note. This has not been done and is not expected to be completed.
Time Frame: from study entry to end of protocol treatment.
Population: T cell responses to tumor cells in vitro have not been analyzed and those analyses are not expected to be completed. Funding ended.
Arm/Group | Group 1: Adjuvant | Group 2: Neoadjuvant
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days after last study intervention, up to 18 months after enrollment.
Description: CTCAE
Arm/Group | Group 1: Adjuvant | Group 2: Neoadjuvant
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Adjuvant (N=3) | Group 2: Neoadjuvant (N=3)
injection site reaction (Skin and subcutaneous tissue disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes